CLINICAL TRIAL: NCT05509309
Title: Promoting Inclusive Educational Environments for Children with Autism and Other Social-communication Challenges: Preschool Class and Primary School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lise Roll-Pettersson, Professor, Stockholm University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VR 2020-03267
Record Dates: First submitted 2022-05-31; First posted 2022-08-22 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder; Social Communication Challenges
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): In the experimental group, in-service training on autism, program quality, and APERS will be provided to participating staff. Furthermore, APERS-rating to assess the program quality for students with ASD/SCC will be conducted. Pertaining feedback on program areas of strength and improvement will be provided by the APERS-raters to the classroom teachers.
  Subsequently, assigned coaches (already employed at the school as special educators or equivalent) will based on the APERS-ratings develop an action plan to improve program quality for students with ASD and SCC, in collaboration with classroom teachers. Subsequently, the coach will provide weekly or bi-weekly coaching to promote program quality during the course of two school semesters (approximately 8-9 months).
  Interventions: Behavioral: APERS-based model
- Comparison group (No Intervention): The classrooms in the comparison group will also be rated with the APERS, and feedback will provided to classroom teachers. However, no further support will be provided in transforming APERS-ratings with pertaining feedback into best practice.

INTERVENTIONS:
Behavioral: APERS-based model — APERS-assessments followed by in-service training, APERS-feedback and on-site coaching to improve primary school classroom quality for students with ASD/SCC
  Arms: Experimental group

SUMMARY:
This study evaluates the effect of using the Autism Program Environment Rating Scale (APERS) as the foundation for providing feedback, in-service training and coaching to teachers, to improve program quality for autistic (ASD) students and students with related social-communication challenges (SCC) in Swedish primary school classrooms. In the current study half of the participating classrooms will receive the APERS-based model for program quality improvement, while the other half will receive services as usual.

It is hypothesized that the APERS-based model will improve primary school program quality for children with ASD and SCC, as well as improve functioning for students with ASD/SCC and self-perceived self-efficacy among participating teachers, compared to the study's comparison group.

ELIGIBILITY:
Inclusion Criteria:

* autism diagnosis
* socio-communicative challenges identified by parents and/or school staff
* attending a primary school classroom (i.e., from pre-school class to third grade)

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in autism program quality assessed with the Autism Program Environment Rating Scale - Preschool and primary school (APERS-Fk/L-SE) | Baseline and about 9 months from baseline
  The APERS-Fk/L-SE is a rating scale designed to examine primary school program quality for autistic students in Sweden. It contains 10 domains including areas such as students' personal independence and competence, and challenging behaviors. The scale consists of 59 items rated on a five-point Likert-scale (1= low quality - 5 = high quality) resulting in individual item scores, subdomain scores, domain scores and a total score.

SECONDARY OUTCOMES:
Change from baseline in how children feel about their school assessed with How I Feel About My School (HIFAMS) | Baseline and approximately 9 months from baseline
  The HIFAMS is a questionnaire designed to assess the happiness and subjective well-being of children in school. It is to to be completed by all children in all participating classrooms in the study. The questionnaire is composed of seven questions which asks children how they feel about school life, which are scored using a three-point Likert "face" scale (sad face, neutral face, happy face).
Change from baseline in parents ratings on their children's body functions, activities and participation and contextual factors assessed with the International Classification of Functioning, Disability and Health (ICF) Core Sets for Autism | Baseline and approximately 9 months from baseline
  the ICF Core Sets for Autism is a questionnaire for parents to complete about their children. It contains a number of statements about their children's body functions, activities and participation, and contextual factors that may affect their children's functioning rater on a Likert-scale from either 0 to 10, or -5 to 5 (contextual factors), where higher ratings indicate higher levels of functioning and participation.
Change from baseline in children's self-regulation and academic behavior assessed with children's self-regulation and academic behavior questionnaire | Baseline and approximately 9 months from baseline
  The Children's self-regulation and academic behavior questionnaire is designed for teachers to rate children's self-regulation and academic behavior skills in various situations in the classroom, rated on a five-point Likert scale from 0 to 4, across 11 items, where higher ratings indicate more skills and better self-regulation.
Change from baseline in teachers' global impression of the child in the classroom | Baseline and approximately 9 months from baseline
  Teachers' global impression of the child in school during the latest week. Rated on a four-point Likert scale from 0 to 3, across four items, where higher ratings indicate more well-being, participation, engagement and adaptive behaviors.
Change in teachers' stress assessed with the Teachers' Stress Scale | Baseline and approximately 9 months from baseline
  The Teachers' Stress Scale is a questionnaire designed for teachers to complete about their perceived work-related stress. It consists of five items, and is rated on a six-point Likert scale from 0 to 6 where higher ratings are associated with more stress.
Change in teachers' perceived self-efficacy for supporting students with autism using the Autism Self-Efficacy Scale for Teachers | Baseline and approximately 9 months from baseline
  The Autism Self-Efficacy Scale for Teachers is a questionnaire for teachers to complete about their perceived self-efficacy for supporting students with ASD and socio-communicative challenges in their classroom. It consists of 28 items, and is rated on a six-point Likert scale from 0 to 5. Higher ratings indicate more self-efficacy.
Change in teachers' work satisfaction assessed with the Teacher Work Satisfaction Questionnaire | Baseline and approximately 9 months from baseline
  The Teacher Work Satisfaction Questionnaire is designed for teachers to complete about their work satisfaction. It contains three items that are rated on a six-point Likert scale from 0 to 5, where higher ratings indicate more work satisfaction,

OTHER OUTCOMES:
Social validity assessed with the Social Validity Scale | Follow-up approximately 9 months after onset of study
  A scale designed to asses the social validity of the procedures, goals and outcomes of the study by participating school staff. It consists of 12 items rated on a Likert scale from 0 to 5, where higher ratings indicate higher levels of perceived social validity.
Social responsiveness measured with the Social Responsiveness Scale 2 (SRS-2) | Baseline assessment
  The SRS-2 is a scale designed to identify the presence and severity of social impairment within the autism spectrum and to differentiate it from that which occurs in other conditions. In the current study used to assess the level of social challenges for the participating "index children" (i.e. children with autism or socio-communicative challenges participating in the study). The scale contains 65 items and is rated by the children's parents. Each item is rated on a scale from 1 to 4, where 1 is "not true" and 4 is "almost always true". Higher scores indicate more severe social impairment associated with autism, while lower scores indicate the opposite.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Pettersson Roll, PhD, Principal Investigator — Stockholm University
Locations (1):
- Stockholm Municipality, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No